CLINICAL TRIAL: NCT06501352
Title: Comparative Study Between Dexmedetomidine & Neostigmine as an Adjuvant to Local Anesthetic Mixture in Peribulbar Block in Vitreoretinal Surgeries
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hussein Hamdy, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Ain Shams University Hospitals
Record Dates: First submitted 2023-01-10; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Vitreoretinal Surgeries; Local Anesthesia
Keywords: Dexmeditomedine; Neostagmine; Peribulbar block
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine; Lidocaine; Hyaluronoglucosaminidase; Neostigmine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmeditomedine group (Active Comparator): Patients in this group will receive Dexmeditomedine in Local anesthesia mixture.
  Interventions: Drug: Dexmedetomidine
- Neostigmine group (Active Comparator): Patients in this group will receive Neostigmine in Local anesthesia mixture.
  Interventions: Drug: Neostigmine
- Control group (Placebo Comparator): Patients in this group will receive saline (placebo) in Local anesthesia mixture.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Additive to Local anesthetic mixture
  Other Names: Marcaine; Xylocaine; Hyaluronidase
  Arms: Dexmeditomedine group
Drug: Neostigmine — Additive to Local anesthetic mixture
  Other Names: Marcaine; Xylocaine; Hyaluronidase
  Arms: Neostigmine group
Drug: Saline — Control
  Other Names: Marcaine; Xylocaine; Hyaluronidase
  Arms: Control group

SUMMARY:
The majority of patients undergoing ophthalmic surgeries are elderly, with multiple chronic diseases, with increased risk of morbidity and mortality under general anesthesia.

Peribulbar anesthesia is widely practiced now as a first-choice local block for ophthalmic surgeries.

Dexmedetomidine is a highly selective alpha-2 adrenoceptor. It increases central and peripheral nerve blockade and when added to local anesthetic as an adjuvant, it will provide better anesthetic quality as well as prolongation of postoperative analgesia .

Neostigmine is a parasympathomimetic drug that increase the level of acetylecholine at peripheral muscarinic receptors present in the peripheral nerve endings .

Many researches examined the analgesic effects of peripherally administered neostigmine as in intravenous regional anesthesia reporting that addition of neostigmine to the local anesthetic solution accelerated the onset of anesthesia

& prolong duration .

DETAILED DESCRIPTION:
81 participants divided into three groups 27 patient in each group with inclusion criteria :

* Patients aged from 21 to 60 years.
* Patients ASA I to II undergoing Vitreoretinal Surgeries.
* Patient with axial globe length below 26 mm.
* Patients consented with Local anesthesia.

The three groups:

group I : will receive Peribulbar anesthesia block via 25G needle is inserted transcutaneously through the inferotemporal approach at the junction between the medial two third and the lateral third of the lower orbital margin in such a way the bevel is facing the globe and the tip towards the floor of the orbit until the needle passes through the orbital septum it is directed then posteriorly tangential to the floor of the orbit for 25mm length at which the 8 ml local anesthetic mixture is injected ( 4 ml of bupivacaine + 3 ml of mixture of Lidocaine & Hyaluronidase +1ml of Dexmedetomidine equivalent to 25 mcg).

Ocular compression is applied for 5 minutes by Honan intraocular pressure IOP reducer adjusted at 20mmHg.

Group II :

Will recieve ( 4 ml of bupivacaine + 3 ml of mixture of Lidocaine & Hyaluronidase +1ml of Neostigmine equivalent to 0.5 mg)

Group III :

( 4 ml of bupivacaine + 3 ml of mixture of Lidocaine & Hyaluronidase +1ml Normal Saline 0.9%)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 21 to 60 years.
* Patients ASA I to II .
* Patient with axial globe length below 26 mm.
* Patients consented with Local anesthesia.

Exclusion Criteria:

* Patient refusal.
* Patients below or above the age.
* Patients with bleeding disorders.
* Patient with axial globe length more than 26 mm.
* history of relevant drug allergy to any of the used drugs

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Onset & Duration of sensory and motor block | 12 hours
  By minutes , Refers to the time from injection till patient will feel nothing in his eyes , then the time when he regain feeling again

SECONDARY OUTCOMES:
Systolic & Diastolic Arterial Blood Pressure | 12 hours
  measuring it pre-operative , intra-operative & post-operative
Heart rate | 12 hours
  measuring HR per minute pre & intra & post operative
Patient & Surgeon satisfaction | 12 hours
  No pain by VAS score ( from 0 to 10 as 0 no pain & 10 maximum pain ) VAS score intraoperative to assess patient satisfaction & surgeon satisfactory by longer duration of motor & sensory block .

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After completion of work
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 month
Access Criteria: husseinhamdy@med.asu.edu.eg